CLINICAL TRIAL: NCT04335942
Title: Characterization of the Postural Habits of Wheelchair Users in an Ecological Situation and Analysis of the Acceptability of International Recommendations in the Prevention of Pressure Sores Risk by Using a Connected Textile Sensor Integrating an Artificial Intelligence Algorithm
Brief Title: Characterization of the Postural Habits of Wheelchair Users Analysis of the Acceptability of International Recommendations in the Prevention of Pressure Sores Risk by Using a Connected Textile Sensor
Acronym: Es-Alert
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP190924
Record Dates: First submitted 2019-11-22; First posted 2020-04-07 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Duchenne Muscular Dystrophy; Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AFNOR 3.6 alerts (Other): Alert called "AFNOR 3.6" in connection with the dispersion index described by Drummond et al 1985 and validated by Sprigle et al 2003. This alert corresponds to the quantification of the percentage of weight on the slick distributed over a small area (55% on one to three zones totalling 30cm2),
  Interventions: Other: Alert "AFNOR 3.6".
- AFNOR 3.6 alerts and Guidelines (Other): AFNOR 3.6" alerts and "Guidelines" alerts. By alertes Guidelines we mean the clinical recommendations of the Spinal Cord medicine association, i.e. weight relief every 15 to 30 minutes (Bergstrom et al., 1992; Nixon, 1985; Ho and Bogie, 2007) over a period of 1 minute 51 (Coggrave and Rose 2003) for spinal cord injuries. For patients who do not push up, a tilt of at least 25° of seat and 120° of backrest or a minimum of 45° in one block (Dicianno et al. 2009).
  Interventions: Other: Alertes " AFNOR 3.6 " et alertes " Guidelines ".

INTERVENTIONS:
Other: Alert "AFNOR 3.6". — This alert corresponds to the quantification of the percentage of weight on the slick distributed over a small area (55% on one to three zones totalling 30cm2),
  Arms: AFNOR 3.6 alerts
Other: Alertes " AFNOR 3.6 " et alertes " Guidelines ". — By alertes Guidelines we mean the clinical recommendations of the Spinal Cord medicine association, i.e. weight relief every 15 to 30 minutes over a period of 1 minute 51 for spinal cord injuries. For patients who do not push up, a tilt of at least 25° of seat and 120° of backrest or a minimum of 45° in one block.
  Arms: AFNOR 3.6 alerts and Guidelines

SUMMARY:
Spinal cord injuries and people with Duchenne Muscular Dystrophy or Infant Spinal Muscular Atrophy (ISA) are prone to pain and pressure sores associated with prolonged sitting. For this reason, it is recommended that people with spinal cord injuries release pressure every 15 to 30 minutes and motorized wheelchair users use the electric positioning functions at least 1 minute every hour.

The aim is to prevent and/or reduce pain and pressure sores. These devices could help to observe daily the variability of users' pressure maps, their impact on occupational performance, the link with pain and redness and could propose customized adjustments.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the impact of an algorithm that characterizes the cruro-ischiatic fingerprints used in daily life and that issues an alert in case of detection of a pressure sore risk defined by the literature on the occupational performance of the subjects.

The resulting assumption is based on the following points:

* The algorithms implemented in this device are able to calculate and isolate a number of cruro-ischiatic fingerprints used during the day during priority activities and active or passive position changes.
* They may, in the event of a risk position, issue alerts based on the recommendations.

This will allow us to analyze the impact of these alerts on the changes in position and relief actually performed by the subject, analyze the consequences on the MCRO score (psychosocial impact on occupational performance) and verify the impact of visual biofeedback on chair positioning.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18 years of age,
* Daily user of a FR (more than 3 hours per day):

  * Persons with Duchenne Muscular Dystrophy (DMD) or DMB using an FRE,
  * People with Infant Spinal Muscular Atrophy (ISA) using an FRE,
  * WB persons using an MRA with sensitivity disorders (ASIA A).
* FRE allowing a switchover of at least:

  * 25° of the seat and 120° of the backrest,
  * 45° of sitting in one block,
* Patient who has signed an informed and written consent,
* Affiliation to a social security scheme (beneficiary or beneficiary).

Exclusion Criteria:

* Refusal of the patient to participate in the study,
* School level lower than cycle 3 not allowing to understand the use of the embedded device,
* Severe incontinence,
* BM without sensitivity disorders,
* Participant in another study or therapeutic trial,
* Patient under guardianship or curatorship,
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the impact of a device, monitoring the wheelchair user's risk of pressure sores and issuing alerts based on international recommendations, on the support reliefs provided by the subject in an ecological situation | 14 days
  Primary outcome will be evaluated with the number of modification of relief or changing of position with or without alert. The metric used will be the number of average reliefs per hour performed by the patient. This number of reliefs will be compared with and without an alert system.

SECONDARY OUTCOMES:
the differences in occupational performance at the MCRO (Mesure canadienne du rendement occupationnel) score | 14 days
  Analyze the differences in occupational performance at the MCRO score. An improvement in MCRO score will mean an improvement of occupational performance in psychosocial dimensions.
the impact of visual biofeedback of the pressure print on chair | 14 days
  Quantify the impact of visual biofeedback of the pressure print on chair positioning by modification of the seat within 5 minutes following the visual cartography consultation
Feasibility study of integrating international recommendations to reduce the risk of pressure ulcers in a medical device | 14 days
  the aim is to verify the technical feasibility of integrating international recommendations to reduce the risk of pressure ulcers in a medical device in relation to the position in the chair through: adequacy between pressure cartography the same label posture over time as well as adequacy between the alert and the type of pressure imprint
the study of the acceptability by the patient of alerts in relation with international recommendations | 14 days
  the study of the acceptability by the patient of alerts in relation with international recommendations will be evaluated with the duration of change in alert characteristics by patient after two days of non-modifiable alerts
the study of the acceptability by the patient of alerts in relation with international recommendations | 14 days
  the study of the acceptability by the patient of alerts in relation with international recommendations will be evaluated with the frequency of change in alert characteristics by patient after two days of non-modifiable alerts

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Hugeron, MD, Principal Investigator — Hôpital Raymond Poincaré
Locations (1):
- Hôpital Raymond Poincaré, Garches, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Drummond D, Breed AL, Narechania R. Relationship of spine deformity and pelvic obliquity on sitting pressure distributions and decubitus ulceration. J Pediatr Orthop. 1985 Jul-Aug;5(4):396-402. doi: 10.1097/01241398-198507000-00002. PMID 3894415
- [Result] Gawlitta D, Li W, Oomens CW, Baaijens FP, Bader DL, Bouten CV. The relative contributions of compression and hypoxia to development of muscle tissue damage: an in vitro study. Ann Biomed Eng. 2007 Feb;35(2):273-84. doi: 10.1007/s10439-006-9222-5. Epub 2006 Nov 29. PMID 17136445
- [Result] Sprigle S, Maurer C, Holowka M. Development of valid and reliable measures of postural stability. J Spinal Cord Med. 2007;30(1):40-9. doi: 10.1080/10790268.2007.11753913. PMID 17385269